CLINICAL TRIAL: NCT00003873
Title: Phase III Trial Comparing a 28 Day Schedule of Daily Oral 5-FU Plus Eniluracil to Protracted Intravenous Infusion in Previously Untreated Patients With Advanced Colorectal Cancer
Brief Title: Fluorouracil With or Without Eniluracil in Treating Patients With Advanced Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02300; E-5296; U10CA021115 (NIH); CDR0000067038 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-07-16 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Adenocarcinoma of the Colon; Adenocarcinoma of the Rectum; Recurrent Colon Cancer; Recurrent Rectal Cancer; Stage IV Colon Cancer; Stage IV Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Fluorouracil; eniluracil

ARMS (2):
- Arm I (Experimental): Patients receive fluorouracil IV as a continuous infusion for 28 days.
  Interventions: Drug: fluorouracil
- Arm II (Experimental): Patients receive eniluracil/fluorouracil orally twice a day for 28 days.
  Interventions: Drug: fluorouracil; Drug: eniluracil

INTERVENTIONS:
Drug: fluorouracil — Given IV or orally
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Drug: eniluracil — Given orally
  Other Names: 776C85; ADH300004; ethynyluracil; GW776; GW776C85
  Arms: Arm II

SUMMARY:
Randomized phase III trial to compare the effectiveness of fluorouracil given by infusion with that of fluorouracil plus eniluracil given by mouth in treating patients who have metastatic, recurrent, or residual advanced colorectal cancer. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known if fluorouracil is more effective with or without eniluracil for advanced colorectal cancer

DETAILED DESCRIPTION:
OBJECTIVES:

I. Compare the response rate, response duration, and survival of patients with advanced colorectal cancer treated with oral fluorouracil (5-FU) and eniluracil or with protracted infusion 5-FU.

II. Compare the toxicity of these treatment regimens in this patient population.

OUTLINE: This is a randomized study. Patients are stratified according to performance status (0 vs 1-2) and measurable disease (yes vs no). Patients are randomized to one of two treatment arms.

ARM I: Patients receive fluorouracil IV as a continuous infusion for 28 days.

ARM II: Patients receive eniluracil/fluorouracil orally twice a day for 28 days.

Treatment continues every 35 days in the absence of disease progression or unacceptable toxicity.

Patients are followed at least every 10 weeks for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with measurable or nonmeasurable histologically confirmed adenocarcinoma of the colon and rectum are eligible provided patient has metastatic, recurrent or residual disease, and tumor is beyond hope of surgical eradication; all pre-study scans documenting disease must be done =< 4 weeks prior to randomization

  * Measurable tumor is defined as a known mass that can be clearly measured in two dimensions by physical examination, CT scan, radionuclide liver scan, or on chest x-ray by a ruler or calipers; the largest diameter of the lesion must measure >= 2 cm by at least one method of evaluation
* Patients must have had no prior therapy for advanced disease
* Patients may have had prior adjuvant treatment with 5-FU provided that the last dose was received > 12 months prior to entering the study; no prior chemotherapy other than adjuvant 5-FU is allowed
* Patients with prior radiotherapy are acceptable, but patients should have measurable or nonmeasurable disease outside the radiation port and/or progressive disease within the previously radiated volume; in addition, it must be at least 2 weeks since administration of radiation therapy and all signs of toxicity must have abated
* Bilirubin =< 1.5 x upper limit of normal (ULN)
* SGOT =< 3 x ULN
* Because Eniluracil changes the metabolism of 5-FU such that it is excreted primarily by the kidneys, an estimated creatinine clearance calculated using the Cockcroft and Gault formula must be obtained in patients with a serum creatinine > institutional normal limits; the estimated creatinine clearance must be >= 50 ml/min prior to starting treatment with Eniluracil/5-FU; if not, a measured creatinine clearance must be done (using a 24 hour urine collection); the measured creatinine clearance must be > 50 ml/min for the patient to be eligible
* Absolute neutrophil count >= 2000 mm³
* Platelet count >= 100,000 mm³
* ECOG performance status 0-2
* No evidence of significant active infection (e.g., pneumonia, peritonitis, wound abscess, etc.) at time of study entry
* No evidence of serious intercurrent illness such as uncontrolled diabetes mellitus, hypothyroidism, malabsorption syndrome or heart failure
* No prior neoplastic diseases (within 5 years) aside from the current malignancy or curatively resected melanoma, skin cancer or cervical carcinoma in situ
* No treatment with folinic acid, interferon, flucytosine or topical 5-FU within the previous 14 days
* Not pregnant or lactating; pregnant and lactating women are excluded from the study because effects on the fetus are unknown and there may be a risk of increased fetal wastage
* Women of childbearing potential and sexually active males are strongly advised to use an accepted and effective method of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 950 (Actual)
Dates: Start 1999-04; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Overall survival | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: John Hines, Principal Investigator — Eastern Cooperative Oncology Group
Locations (1):
- Eastern Cooperative Oncology Group, Boston, Massachusetts, United States